CLINICAL TRIAL: NCT00037336
Title: Atherosclerosis in Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: Vanderbilt University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, C. Michael Stein, Professor of Medicine, Vanderbilt University
Other Study IDs: 1163; R01HL067964 (NIH)
Record Dates: First submitted 2002-05-16; First posted 2002-05-17 (Estimated); Last update posted 2014-03-17 (Estimated); Status verified 2014-03

CONDITIONS: Atherosclerosis; Cardiovascular Diseases; Heart Diseases; Inflammation; Arthritis, Rheumatoid
MeSH Terms: conditions — Atherosclerosis; Cardiovascular Diseases; Heart Diseases; Inflammation; Arthritis, Rheumatoid

SUMMARY:
To test the theory that accelerated inflammation-promoted atherosclerosis occurs in patients with rheumatoid arthritis (RA).

DETAILED DESCRIPTION:
BACKGROUND:

Premature cardiovascular disease is a major cause of mortality in rheumatoid arthritis (RA). The mechanisms underlying accelerated atherosclerosis and its relationship to inflammation in RA are poorly understood. Recent studies indicate that inflammation through the effects of inflammatory cytokines, and oxidative stress, through lipid peroxidation, are important in the pathogenesis of atherosclerosis. The study's hypothesis is that accelerated, inflammation-promoted atherosclerosis occurs in RA.

DESIGN NARRATIVE:

The study tests the hypotheses: 1) that structural and functional vascular damage is more frequent and more severe in patients with established RA than matched controls and is related to cumulative disease severity; 2) that this impairment of vascular integrity is associated with clinical and laboratory markers of inflammation, plasma homocysteine concentrations, and oxidative stress. To address these two hypotheses the relationship between longstanding inflammation and vascular integrity will be determined in a cross-sectional study of 75 patients with established RA in whom prospectively obtained clinical data are available for 15 years, and 75 matched non-RA controls. Endothelium-dependent, flow-mediated dilation of the brachial artery measured by ultrasound, and coronary calcium volume measured by electron beam computed tomography (EBCT) will provide functional and structural measures of vascular integrity, respectively. F2-isoprostane excretion, a reliable index of lipid peroxidation in vivo, homocysteine and lipid concentrations will be measured. Vascular integrity, oxidative stress, lipids and homocysteine will be compared in controls and RA patients. In the RA patients the relationship between RA activity and damage indices obtained over 15 years and vascular function and damage measures will be determined. Using the same techniques we will address hypothesis 3) that the rate of progression of vascular disease in patients with early RA can be altered by control of inflammation. In a prospective cohort of 100 patients with early RA receiving usual clinical care and 100 matched non-RA controls followed over 24 months the relationship between clinical and biochemical measures of inflammation and vascular integrity will be determined by comparing "responders" and "non-responders". These studies will provide a basic understanding of the interrelationship between inflammation, lipids, oxidative stress and vascular damage, and will suggest strategies for reversing or preventing such damage in RA and, potentially, other diseases.

ELIGIBILITY:
must meet ACR criteria for RA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: people with rheumatoid arthritis
Dates: Start 2001-09; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Stein, Principal Investigator — Vanderbilt University

REFERENCES:
- [Background] Sokka T, Pincus T. Eligibility of patients in routine care for major clinical trials of anti-tumor necrosis factor alpha agents in rheumatoid arthritis. Arthritis Rheum. 2003 Feb;48(2):313-8. doi: 10.1002/art.10817. PMID 12571838
- [Background] Sokka T, Pincus T. Contemporary disease modifying antirheumatic drugs (DMARD) in patients with recent onset rheumatoid arthritis in a US private practice: methotrexate as the anchor drug in 90% and new DMARD in 30% of patients. J Rheumatol. 2002 Dec;29(12):2521-4. PMID 12465145
- [Background] Sokka T, Pincus T. Most patients receiving routine care for rheumatoid arthritis in 2001 did not meet inclusion criteria for most recent clinical trials or american college of rheumatology criteria for remission. J Rheumatol. 2003 Jun;30(6):1138-46. PMID 12784382
- [Background] Olsen NJ, Stein CM. New drugs for rheumatoid arthritis. N Engl J Med. 2004 May 20;350(21):2167-79. doi: 10.1056/NEJMra032906. No abstract available. PMID 15152062
- [Background] Pincus T, Yazici Y, Sokka T, Aletaha D, Smolen JS. Methotrexate as the "anchor drug" for the treatment of early rheumatoid arthritis. Clin Exp Rheumatol. 2003 Sep-Oct;21(5 Suppl 31):S179-85. PMID 14969073
- [Background] Sokka T, Willoughby J, Yazici Y, Pincus T. Databases of patients with early rheumatoid arthritis in the USA. Clin Exp Rheumatol. 2003 Sep-Oct;21(5 Suppl 31):S146-53. PMID 14969067
- [Background] Pincus T, Sokka T. Uniform databases in early arthritis: specific measures to complement classification criteria and indices of clinical change. Clin Exp Rheumatol. 2003 Sep-Oct;21(5 Suppl 31):S79-88. PMID 14969056
- [Background] Olsen N, Sokka T, Seehorn CL, Kraft B, Maas K, Moore J, Aune TM. A gene expression signature for recent onset rheumatoid arthritis in peripheral blood mononuclear cells. Ann Rheum Dis. 2004 Nov;63(11):1387-92. doi: 10.1136/ard.2003.017194. PMID 15479887
- [Background] Pincus T, Sokka T, Kautiainen H. Patients seen for standard rheumatoid arthritis care have significantly better articular, radiographic, laboratory, and functional status in 2000 than in 1985. Arthritis Rheum. 2005 Apr;52(4):1009-19. doi: 10.1002/art.20941. PMID 15818706
- [Background] Yazici Y, Sokka T, Kautiainen H, Swearingen C, Kulman I, Pincus T. Long term safety of methotrexate in routine clinical care: discontinuation is unusual and rarely the result of laboratory abnormalities. Ann Rheum Dis. 2005 Feb;64(2):207-11. doi: 10.1136/ard.2004.023408. Epub 2004 Jun 18. PMID 15208176
- [Background] Sokka T, Pincus T. An Early Rheumatoid Arthritis Treatment Evaluation Registry (ERATER) in the United States. Clin Exp Rheumatol. 2005 Sep-Oct;23(5 Suppl 39):S178-81. PMID 16273804
- [Background] Chung CP, Oeser A, Raggi P, Gebretsadik T, Shintani AK, Sokka T, Pincus T, Avalos I, Stein CM. Increased coronary-artery atherosclerosis in rheumatoid arthritis: relationship to disease duration and cardiovascular risk factors. Arthritis Rheum. 2005 Oct;52(10):3045-53. doi: 10.1002/art.21288. PMID 16200609
- [Background] Asanuma Y, Xie HG, Stein CM. Pharmacogenetics and rheumatology: Molecular mechanisms contributing to variability in drug response. Arthritis Rheum. 2005 May;52(5):1349-59. doi: 10.1002/art.21027. No abstract available. PMID 15880820